CLINICAL TRIAL: NCT02168127
Title: A Six-month, Open-label, Multi-center Study of the Safety and Efficacy of PRC-063 in Adults and Adolescents With ADHD
Brief Title: Long-Term Safety of PRC-063 in Adolescents and Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 063-012
Record Dates: First submitted 2014-06-14; First posted 2014-06-20 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active drug group (Experimental): PRC-063 - Active methylphenidate hydrochloride extended-release capsules drug group
  Interventions: Drug: Drug: PRC-063; Drug: PRC-063

INTERVENTIONS:
Drug: Drug: PRC-063 — Methylphenidate Hydrochloride Extended-Release Capsules
  Other Names: Methylphenidate
Drug: PRC-063 — Methylphenidate Hydrochloride Extended-Release Capsules
  Other Names: Methylphenidate

SUMMARY:
The purpose of this six month, open-label study is to evaluate the long-term safety and efficacy of PRC-063 in adults and adolescents with ADHD.

DETAILED DESCRIPTION:
This is an open label, multicenter, phase 3 study to evaluate the safety and efficacy of PRC-063 (methylphenidate hydrochloride controlled-release capsules 25, 35, 45, 55, 70, 85 or 100 mg/day) in the treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in adolescent subjects aged ≥12 to <18 years of age and adult subjects aged ≥18 years of age. In order to participate, subjects must have completed Purdue Pharma Study 063-009 or Purdue Pharma Study 063-010. This study will be conducted at approximately 50 centers across the United States and Canada. After giving written informed consent (as well as informed assent for subjects <18 years of age), subjects will be screened to ascertain their suitability for the study according to the inclusion and exclusion criteria. There will be seven monthly efficacy and safety visits during which subjects will be assessed on active, open-label PRC-063. The starting dose will be at the discretion of the Investigator. Dose-adjustment visits may occur weekly to optimize the subject's dose via titration. For adolescent subjects, the maximum dose will be 85 mg/day. For adult subjects, the maximum dose will be 100 mg/day.

ELIGIBILITY:
Inclusion Criteria: Subjects must satisfy the following criteria to be enrolled in the study as an adolescent:

• Male or non-pregnant, non-nursing female at least 12 years of age and less than 18 years of age.

Subjects must satisfy the following criteria to be enrolled in the study as an adult:

• Male or non-pregnant, non-nursing female at least 18 years of age and meeting the local, legal definition of adult.

All subjects must also satisfy the following criteria to be enrolled in the study:

* Confirmation of ADHD diagnosis made at Visit 1 of Study 063-009 or 063-010 (inattentive, hyperactive/impulsive or combined-type, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition based on clinician assessment using multiple informants and a structured interview).
* Female subjects must be one of the following:
* Surgically sterile prior to screening
* Postmenopausal
* if of childbearing potential, abstinent or willing to use a reliable method of contraception, such as oral contraceptive, two barrier methods, a barrier method plus a spermicidal agent.
* Female subjects of Child-Bearing Potential (FOCP) must have a negative serum β-hCG pregnancy test, as assessed at Visit 6 of Study 063-009 or 063-010 (data will not be available at the time of entry).
* If the subject is an adult, mentally and physically competent to sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study. If the subject is an adolescent, mentally and physically competent to sign an informed assent document, in the case of the subject, and an informed consent document, in the case of the parent/guardian, indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Able and willing to comply with the study procedures for the entire length of the study.

Exclusion Criteria:

* • Having met any exclusion criteria for Study 063-009 or 063-010.

  * Having been diagnosed during Study 063-009 or 063-010 with strokes, epilepsy, migraine headaches (greater than 1 instance every two months), glaucoma, thyrotoxicosis, tachyarrhythmias or severe angina pectoris or have serious or unstable medical illness. Subjects with controlled or stable asthma or diabetes will be permitted.
  * Elevated blood pressure, defined as any values above 89 diastolic or 139 systolic, as assessed at Visit 6 of Study 063-009 or 063-010.
  * Clinically significant ECG abnormalities, as assessed at Visit 6 of Study 063-009 or 063-010 (data will not be available at the time of entry).
  * Clinically significant laboratory abnormalities, as assessed at Visit 6 of Study 063-009 or 063-010 (data will not be available at the time of entry).
  * Currently receiving guanethidine, pressor agents, MAO inhibitors, coumarin anticoagulants, anticonvulsants (e.g. phenobarbital, phenytoin, primidone), phenylbutazone, tricyclic antidepressants (e.g. imipramine, desipramine), selective serotonin reuptake inhibitors (SSRIs) or herbal remedies (unless on a stable dose for 4 weeks).
  * If the Investigator judges that continued treatment with PRC-063 is not in the subject's best interest.
  * Subjects who are currently considered a suicide risk by the investigator.
  * Having been diagnosed during Study 063-009 or 063-010 with schizophrenia, schizoaffective disorder, primary affective disorder, schizotypal personality, major depression, bipolar disorder, generalized anxiety, borderline personality disorder, antisocial personality or another unstable psychiatric condition requiring treatment.
  * Having been diagnosed during Study 063-009 or 063-010 with physiological dependence (excluding nicotine) on narcotic analgesics or other psychoactive drugs (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines).
  * Excessive consumption of alcohol occurring during Study 063-009 or 063-010 (consumes alcohol in quantities greater than 15 drinks per week on average; 1 drink is defined as 360 mL/12 oz. of beer, 120 mL/4 oz. of wine, or 30 mL/1 oz. of hard liquor).
  * Currently (or within 30 days before the planned start of treatment) receiving an investigational drug or using an experimental medical device, other than PRC-063.
  * Homeless.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
occurrence of treatment-emergent adverse events | Within 6 months

SECONDARY OUTCOMES:
Clinician-administered ADHD-5-Rating Scale | Within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Reiz, Study Director — Purdue Pharma LP
Locations (35):
- United States (30):
  - UCLA, Los Angeles, California
  - Synergy Clinical Research, National City, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Orange County Neuro Phychiatry Research Centre, Orange, California
  - Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Research, Gainesville, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - CNS Healthcare Jacksonville, Jacksonville, Florida
  - Florida Clinical Research Center, Maitlin, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Advanced Clinical Research, Boise, Idaho
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Medical Research Network, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigation, Portland, Oregon
  - Oregon Center for Clinical Investigation, Salem, Oregon
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Houston Clinical Trials, Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Ericksen Research, Clinton, Utah
  - Physiciatric and Behavioral Solutions, Salt Lake City, Utah
  - Woodstock Research Center at Neuropsychiatric Associates, Woodstock, Vermont
  - NeuroScience, Herndon, Virginia
  - Northwest Clinical Research Center, Friday Harbor, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
- Canada (5):
  - Dr. Margaret Weiss, Vancouver, British Columbia
  - Doctors Jackiewicz Professional Medical Corporation, Niagara Falls, Ontario
  - Dr. Judy van Stralen, Ottawa, Ontario
  - The Kids Clinic, Whitby, Ontario
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- [Derived] Weiss MD, Surman C, Khullar A, Owens J, He E, Cataldo M, Donnelly G. Effect of a Multilayer, Extended-Release Methylphenidate Formulation (PRC-063) on Sleep in Adolescents with Attention-Deficit/Hyperactivity Disorder: A Randomized, Double-Blind, Fixed-Dose, Placebo-Controlled Trial Followed by a 6-Month Open-Label Follow-Up. J Child Adolesc Psychopharmacol. 2021 Nov;31(9):623-630. doi: 10.1089/cap.2021.0087. Epub 2021 Oct 28. PMID 34714112
- [Derived] Weiss MD, Cutler AJ, Kollins SH, Donnelly GAE. Efficacy and Safety of a Long-Acting Multilayer-Release Methylphenidate Formulation (PRC-063) in the Treatment of Adolescent Attention-Deficit/Hyperactivity Disorder: A Randomized, Double-Blind Clinical Trial with a 6-Month Open-Label Extension. J Child Adolesc Psychopharmacol. 2021 Nov;31(9):610-622. doi: 10.1089/cap.2021.0034. Epub 2021 Oct 8. PMID 34637343
- [Derived] Weiss MD, Surman C, Khullar A, He E, Cataldo M, Donnelly G. Effect of a Multi-Layer, Extended-Release Methylphenidate Formulation (PRC-063) on Sleep in Adults with ADHD: A Randomized, Double-Blind, Forced-Dose, Placebo-Controlled Trial Followed by a 6-month Open-Label Extension. CNS Drugs. 2021 Jun;35(6):667-679. doi: 10.1007/s40263-021-00814-z. Epub 2021 May 31. PMID 34057707